CLINICAL TRIAL: NCT04595695
Title: The Effect of Clear Masks in Improving Patient Relationships
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20-2229
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-10

CONDITIONS: Communication; Trust; Covid19; Surgery
Keywords: Masks
MeSH Terms: conditions — Communication; COVID-19

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into typical covered mask versus transparent mask worn by the surgeon.
Who Masked: Participant
Masking Description: Patients will not know that their surgeon is participating in a research study. Visits will be completed as they typically would with the surgeon wearing a mask.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transparent Mask (Experimental): Surgeons will be provided a transparent mask for use during in-person clinic visits with a new patient. Otherwise, visits will be conducted as per usual and the patient will be surveyed immediately after the visit.
  Interventions: Behavioral: Transparent mask
- Covered Mask (Active Comparator): Surgeons will be instructed to wear a typical, covered mask for the in-person clinic visit with a new patient. The visit will be conducted as it typically would, and the patient will be surveyed immediately after the visit.
  Interventions: Behavioral: Typical surgical covered mask

INTERVENTIONS:
Behavioral: Transparent mask — A transparent mask worn by the surgeons in customary fashion will be used.
  Other Names: ClearMask
  Arms: Transparent Mask
Behavioral: Typical surgical covered mask — A standard covered surgical mask worn by the surgeons in in customary fashion will be used.
  Other Names: Halyard
  Arms: Covered Mask

SUMMARY:
To evaluate the effect of wearing masks that hide a surgeon's facial features versus one that shows them. New patients with no prior relationship with the surgeon will be asked questions regarding communication and trust with the surgeon.

DETAILED DESCRIPTION:
Surgeons within the University of North Carolina Department of Surgery will be recruited via an email list-serve. This recruitment email will describe the study and have the consent attached. If the surgeons are interested in participating they will respond to the email and sign the consent form.

The project personnel will arrange to attend their clinic that has new patients scheduled. A random group generator will be used to randomize the patients. The surgeons will be provided either a transparent mask that demonstrates their full facial features or their typical mask that covers their mouth, for each new patient visit. Following each visit, the surgeon will tell the project personnel that they are complete and the project personnel will enter the room, introduce the project, obtain verbal consent (enroll the patient) and if agreeable, provide a brief verbal survey to the patient. The survey will entail confidential questions regarding basic demographics, surgeon communication and trust, as well as an impression of the masks. Survey answers will be Likert scale and open ended. Patients will also be given a debriefing form at the completion of their participation. Surgeons will be asked their impression of the mask at the completion of their participation. All data will be kept confidential on password protected devices.

If patients do not agree to the study they will not be included. If surgeons feel uncomfortable at any point they may withdraw from the study. Any patient demonstrating concerning symptoms of an infection will not be included in the study.

The investigators expect to recruit 10 surgeons, with 10 patients each, totally 100 patients (50 in each arm, clear vs. covered mask). Using Mann-Whitney U test, data will be analyzed for differences in responses between the two groups. Demographic data for both the patient and surgeon will also be analyzed. Patient comments will be qualitatively analyzed for themes by trained researchers.

ELIGIBILITY:
Inclusion Criteria Surgeon:

* Faculty within Department of Surgery at the University of North Carolina at Chapel Hill
* Must be English speaking
* Plans to see new in person visits in clinic

Exclusion Criteria Surgeon:

* None

Inclusion Criteria Patient:

* At least 18 years old
* Can understand and speak English without the use of an interpreter
* Has capacity to make independent medical decisions

Exclusion Criteria Surgeon:

* Has a prior relationship with the surgeon
* Has symptoms of a respiratory infection (cough, shortness of breath, fever)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Patient Mask Preference Quantitative | During 1-minute survey assessed immediately after clinic visit completion
  Using a Likert scale question evaluating patient preference for the type of mask (What was your impression of the surgeon's mask? "Did not like the mask", "somewhat did not like the mask", "somewhat liked the mask", "completely liked the mask", scored as 1 to 4 with higher score indicating greater preference).
Patient Mask Preference Qualitative | During 1-minute survey assessed immediately after clinic visit completion
  Patients will be asked for their comments about the surgeon's mask and these will be immediately transcribed.
Patient Survey Scores Evaluating Surgeon Communication Skills | During 1-minute survey assessed immediately after clinic visit completion
  Using Likert scale questions evaluating patient perception of surgeon communication, taken from the Clinician and Group Consumer Assessment of Healthcare Providers and Systems (CG-CAHPS) healthcare survey, each scored 1-4 with higher number indicating greater communication skills, from "not at all", "somewhat", "mostly" to "completely". This will include 6 questions evaluating communication skills with identical answer choices. Each participants total score will range from 6 to 24 with higher indicating better communication skills.
Patient Survey Scores Describing Trust in the Surgeon | During 1-minute survey assessed immediately after clinic visit completion
  Using Likert scale questions evaluating patient trust of the surgeon, asked, "How comfortable do you feel trusting this surgeon's decisions". Answer choices are score 1 - 4 with 4 indicating great trust, from "Completing uncomfortable", "somewhat uncomfortable", "somewhat comfortable", "completely comfortable"

CONTACTS AND LOCATIONS:
Overall Officials: Ian Kratzke, MD, Principal Investigator — University of North Carolina at Chapel Hill Department of Surgery
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Surgeon-identifying information will only be available to the primary investigator and will not be shared. Patient-identifying information will not be collected beyond basic demographics. Patient quotations may be published but will not be identifiable.

REFERENCES:
- [Derived] Kratzke IM, Rosenbaum ME, Cox C, Ollila DW, Kapadia MR. Effect of Clear vs Standard Covered Masks on Communication With Patients During Surgical Clinic Encounters: A Randomized Clinical Trial. JAMA Surg. 2021 Apr 1;156(4):372-378. doi: 10.1001/jamasurg.2021.0836. PMID 33704389